CLINICAL TRIAL: NCT00455520
Title: A Randomized-Withdrawal Phase 3 Study Evaluating the Safety and Efficacy of CG5503 Extended Release (ER) in Subjects With Painful Diabetic Peripheral Neuropathy
Brief Title: A Safety and Efficacy Study for Tapentadol (CG5503) Extended Release for Patients With Painful Diabetic Peripheral Neuropathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR012466; R33133PAI3015 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.)
Record Dates: First submitted 2007-04-01; First posted 2007-04-03 (Estimated); Results first posted 2010-01-13 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Diabetic Neuropathy
Keywords: Diabetic neuropathy; Painful Diabetic Polyneuropathy; Polyneuropathy; Peripheral neuropathy
MeSH Terms: conditions — Diabetic Neuropathies; Polyneuropathies; Peripheral Nervous System Diseases | interventions — Tapentadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): placebo matching placebo twice daily for 12 weeks
  Interventions: Drug: placebo
- CG5503 (Experimental): CG5503 100, 150, 200, 250mg twice daily given for up to 15 weeks
  Interventions: Drug: CG5503

INTERVENTIONS:
Drug: CG5503 — 100, 150, 200, 250 mg twice daily given for up to 15 weeks
  Arms: CG5503
Drug: placebo — matching placebo twice daily for 12 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effectiveness (level of pain control) and safety of Tapentadol (CG5503) extended release (ER) (base) compared to placebo in patients with moderate to severe pain from diabetic peripheral neuropathy.

DETAILED DESCRIPTION:
The primary objective of this randomized-withdrawal (randomized means study medication assigned to patients by chance and withdrawal means to stop using), multicenter, double-blind (neither patient nor investigator knows the study medication), placebo-controlled, Phase 3 study is to determine the effectiveness and safety of orally administrated Tapentadol (CG5503) extended release (ER) (base) at doses of 100-250 mg twice daily in patients with moderate to severe pain from diabetic peripheral neuropathy. The study is being conducted for registration and approval of CG5503 in the US and outside US. The trial will consist of two phases: Phase I is open-label and Phase 2 is double- blind. In the Open-Label Phase 1 there will be four periods: screening (to assess eligibility), washout (dependent on the pain medication the patient was previously taking), pain intensity perctoris evaluation (over a 3 day period), and open-label titration (study drug will be titrated to an optimal dose starting with 50 mg twice a day and adjusted to an optimal dose for a period of 3 weeks). Patients with at least a 1-point reduction in the average pain intensity score at the end of the open-label titration period, as compared with pre-titration will be eligible for randomization in the double-blind phase. In the double-blind Phase 2, there will be two periods: double-blind maintenance period (take drug for 12 weeks), and follow-up (a visit within 4 days of the intake of the last dose of study drug and a follow-up call approximately 10-14 days after the intake of the last dose of the study drug). The patient will maintain the dose level achieved at the end of the Phase 1 during the double-blind treatment phase. The study hypothesis is that the study drug will be different from placebo in the change in pain intensity. Titrate Tapentadol (CG5503) extended release (ER) 50 mg to patient's optimal dose ranging between 100mg and 250mg twice a day; Placebo (no active ingredients). All doses of trial treatment will be taken orally with or without food, for a maximum timeframe of 15 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 1 or Type 2 diabetes mellitus must have a documented clinical diagnosis of painful diabetic peripheral neuropathy with symptoms and signs for at least 6 months, and pain present at the time of screening
* The investigator considers the patient's blood glucose to be controlled by diet, or hypoglycemics, or insulin for at least 3 months prior to enrolling in the study (this control should be documented by figures of glycated hemoglobin [HbA1c] no greater than 11% at screening)
* Patients have been taking analgesic medications for the condition for at least 3 months prior to screening (patients taking opioid analgesics must be dissatisfied with current treatment, and patients taking non-opioid analgesics must be dissatisfied with current analgesia)
* Patients currently requiring opioid treatment must be taking daily doses of an opioid-based analgesic equivalent to <=160 mg of oral morphine

Exclusion Criteria:

* No significant pulmonary, gastrointestinal, endocrine, metabolic (except diabetes mellitus), neurological, psychiatric disorders (resulting in disorientation, memory impairment or inability to report accurately as in schizophrenia, Alzheimer's disease), or any other clinically significant disease that in the Investigator's opinion may affect efficacy or safety assessments or may compromise patient's safety during trial participation
* no history of moderate to severe hepatic impairment such as chronic hepatitis B or C, presence of active hepatitis B or C within the last 3 months or impaired hepatic function with ALT or AST greater than 3-fold ULN
* No patients with severely impaired renal function
* No laboratory values above or below limits of normal unless considered not clinically relevant by the Investigator
* No significant cardiac disease (e.g., unstable angina pectoris, angina pectoris Canadian Cardiovascular Society (CCS) class III-IV, acute myocardial infarction within the last 3 months, cardiac insufficiency New York Heart Association (NYHA) class III-IV) or significant vascular disease (e.g., peripheral arterial occlusive disease (PAOD) Fontaine class IIb-IV)
* no life-long history of seizure disorders or epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 395 (Actual)
Dates: Start 2007-04; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Afilalo M, Morlion B. Efficacy of tapentadol ER for managing moderate to severe chronic pain. Pain Physician. 2013 Jan;16(1):27-40. PMID 23340531
- [Derived] Schwartz S, Etropolski M, Shapiro DY, Okamoto A, Lange R, Haeussler J, Rauschkolb C. Safety and efficacy of tapentadol ER in patients with painful diabetic peripheral neuropathy: results of a randomized-withdrawal, placebo-controlled trial. Curr Med Res Opin. 2011 Jan;27(1):151-62. doi: 10.1185/03007995.2010.537589. PMID 21162697

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period for this out-patient, multicenter study occurred between 15 March 2007 and 20 August 2008.
Pre-assignment Details: The study consisted of a 2-week screening period followed by a 3-week open-label phase where all subjects received tapentadol extended release (ER) and were titrated to an optimal dose, and a 12-week double-blind phase where subjects were randomly assigned to receive tapentadol ER or placebo.
Groups:
- Tapentadol ER: Tapentadol ER dose of 100 to 250mg twice a day (BID) for 12 weeks during the double blind period. The study medication was provided as tablets taken orally.
- Placebo: Placebo tablets taken orally twice a day (BID) for 12 weeks during the double blind period.
Period: Open Label Tapentadol Extended Release
Arm/Group | Tapentadol ER | Placebo
Started | 591 | 0
Completed | 395 | 0
Not Completed | 196 | 0
Not completed — Withdrawal by Subject | 24 | 0
Not completed — Lost to Follow-up | 3 | 0
Not completed — Adverse Event | 100 | 0
Not completed — Lack of Efficacy | 23 | 0
Not completed — Study drug non-compliant | 13 | 0
Not completed — All other | 33 | 0
Period: Double Blind Tapentadol ER vs Placebo
Arm/Group | Tapentadol ER | Placebo
Started | 196 (2 subjects enrolled two separate times in this study, 1 subject did not receive study medication) | 193 (1 subject enrolled two separate times in this study, 2 subjects did not receive study medication)
Completed | 133 | 131
Not Completed | 63 | 62
Not completed — Adverse Event | 29 | 15
Not completed — Lack of Efficacy | 8 | 29
Not completed — Withdrawal by Subject | 15 | 7
Not completed — Lost to Follow-up | 3 | 3
Not completed — Study drug non compliant | 4 | 2
Not completed — All other | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tapentadol ER | Placebo | Total
Number analyzed (Participants) | 196 | 193 | 389
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 136 | 120 | 256
  >=65 years | 60 | 73 | 133
Age Continuous [Mean (Standard Deviation); unit: years] | 59.9 (10.68) | 60.6 (10.56) | 60.2 (10.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 77 | 154
  Male | 119 | 116 | 235
Region of Enrollment [Number; unit: participants]
  United States | 191 | 189 | 380
  Canada | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (at Randomization) in Average Pain Intensity on an 11-point Numerical Rating Scale (NRS) Over the Last Week of the Double-blind Maintenance Period at Week 12
Description: For this twice daily pain assessment, the subjects were to indicate the level of pain experienced over the previous 12 hours on an 11-point Numerical Rating Scale (NRS) where a score of 0 indicated "no pain" and a score of 10 indicated "pain as bad as you can imagine".
Time Frame: Baseline and 12 weeks
Population: Intent to Treat (ITT) analysis set included all randomized subjects who took at least one dose of study medication during the double blind maintenance period with the exception of 3 subjects who were enrolled in the study twice.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Tapentadol ER | Placebo
Number analyzed (Participants) | 196 | 192
scores on a scale | -0.1 (1.69) | 1.3 (2.41)
Statistical Analysis 1: Comparison: Tapentadol ER vs Placebo; Analysis of Covariance Model with factors of treatment, country, prior opioid use, and baseline dose level and start of DB pain score as factors; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -1.3, 95% CI [-1.7 to -0.92], Standard Error of Mean 0.20

2. Secondary Outcome: The Number of Patients Achieving at Least 30% Improvement in Pain Score at Week 12 of the Double-blind Maintenance Period From the Start of the Open Label Period.
Description: The number of patients achieving at least 30% improvement in pain score at Week 12 of the double-blind maintenance period on an 11-point numerical rating scale compared with the start of the open-label period.
Time Frame: Start of Open Label and at 12 weeks of Double Blind
Population: Intent-to-treat analysis set.
Measure: Number; unit: participants
Arm/Group | Tapentadol ER | Placebo
Number analyzed (Participants) | 196 | 192
participants | 105 | 81

3. Secondary Outcome: Percentage of Patients Who Reported Very Much Improved or Much Improved From Baseline in Patient Global Impression of Change Over the Last Week of the Maintenance Period at Week 12
Description: Percentage of patients who reported very much improved (1) or much improved (2) based on an ordinal measure indicating change from start of double blind treatment (on a scale of 7 = Very much worse to 1 = Very much improved)
Time Frame: 12 week endpoint
Population: as for outcome 1
Measure: Number; unit: percentage of patients
Arm/Group | Tapentadol ER | Placebo
Number analyzed (Participants) | 177 | 180
percentage of patients | 64 | 38

4. Secondary Outcome: Change From Baseline in EuroQol-5 (EQ-5D) Health Status Index to Week 12
Description: Change from baseline to end point in EuroQol-5 Dimension Questionnaire. A higher score indicates an improvement in health in the Health Status Index. The EuroQol-5 is a five dimensional health state classification. Each dimension is assessed on a 3-point ordinal scale (1=no problems, 2=some problems, 3=extreme problems). The responses to the five EQ-5D dimensions were scored using a utility-weighted algorithm to derive an EQ-5D health status index score between 0 to 1, with 1.00 indicating "full health" and 0 representing dead.
Time Frame: 12 week endpoint (change from baseline)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Tapentadol ER | Placebo
Number analyzed (Participants) | 195 | 192
scores on a scale | 0.7 (0.21) | 0.6 (0.26)

5. Secondary Outcome: Change From Baseline in Sleep Latency Time in Hours Over the Last Week of the Maintenance Period at Week 12.
Description: A Sleep Questionnaire addressed the following question: "How long after bedtime/lights out did you fall asleep last night (hours)?" 12 week endpoint-mean changes from baseline at endpoint for sleep latency. Decrease in time (hours) indicates improvement.
Time Frame: Baseline and 12 week endpoint
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Tapentadol ER | Placebo
Number analyzed (Participants) | 133 | 143
Hours | -0.2 (3.22) | -0.59 (2.77)

6. Secondary Outcome: Change From Baseline in Brief Pain Inventory (BPI) Total Pain Score Over the Last Week of the Maintenance Period at Week 12.
Description: Total pain score where zero equals "no pain" to ten equals "pain as bad as you can imagine" from 12 week endpoint vs baseline.
Time Frame: Baseline and12 week endpoint
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Tapentadol ER | Placebo
Number analyzed (Participants) | 194 | 192
Scores on a scale | -3.1 (2.13) | -2.2 (2.17)

ADVERSE EVENTS:
Time Frame: All adverse events were reported from the time a signed and dated informed consent was obtained throughout the follow-up phase of the study. Serious adverse events were collected for 30 days after the last dose of study drug.
Arm/Group | Tapentadol ER | Placebo
Serious Adverse Events (participants affected / at risk) | 10/196 | 3/193
Other Adverse Events (participants affected / at risk) | 87/196 | 48/193
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tapentadol ER (N=196) | Placebo (N=193)
Helicobacter gastritis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Prostate infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Blood glucose increased (Investigations) | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tapentadol ER (N=196) | Placebo (N=193)
Nausea (Gastrointestinal disorders) | 27 | 12
Diarrhoea (Gastrointestinal disorders) | 16 | 8
Vomiting (Gastrointestinal disorders) | 13 | 2
Constipation (Gastrointestinal disorders) | 12 | 2
Dizziness (Nervous system disorders) | 15 | 3
Headache (Nervous system disorders) | 10 | 10
Anxiety (Psychiatric disorders) | 18 | 8
Restlessness (Psychiatric disorders) | 11 | 8
Insomnia (Psychiatric disorders) | 10 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 13 | 14
Bone pain (Musculoskeletal and connective tissue disorders) | 8 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication. The sponsor can embargo for an additional 60 days to allow for the filing of a patent application.